CLINICAL TRIAL: NCT00245687
Title: A Comparative Study of the Tiger Tube Frictional Nasal Jejunal Feeding Tube and the Dubhoff Tube
Brief Title: A Research Study to Test (2) Two Different Types of Feeding Tubes Used in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05U.229
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: no Primary Disease; ICU Patient Who Require Enteral Nutrition
Keywords: feeding tube, nutrition, gastric, jejunal

INTERVENTIONS:
Device: Tiger Tube

SUMMARY:
The purpose of this study is to compare the success rates of two types of feeding tubes, specifically the standard gastric feeding tube to a small bowel feeding tube.

DETAILED DESCRIPTION:
Enteral nutrition has many advantages for critically ill patients including lower incidence of infections and a reduced hospital stay, however it is controversial whether enteral feeding via small bowel feeding tubes offers an advantage over gastric feeding tubes in terms of reducing aspiration risk, improving feeding tolerance or ensuring quicker attainment of nutritional goals. The advantages of a small bowel feeding tube over a gastric feeding tube is thought to be related to its post pyloric position, however the insertion of small bowel feeding tubes is technically challenging (most studies report a success rate of 15-30%), can take time and has complications not unlike those of the gastric feeding tube. Our hypothesis is that the small bowel feeding tube offers an advantage to the gastric feeding tube due to its ability to achieve post pyloric placement. Specifically we chose to compare the standard gastric feeding tube (Dubhoff) to a small bowel feeding tube which offers the advantage of having alternating flaps which allows the gut to drag this tube into the small bowel.

ELIGIBILITY:
Inclusion Criteria:

* all ICU patients requiring enteral nutrition

Exclusion Criteria:

* coagulopathy, esophageal or gastric, surgery, varices, trauma, ulcer, structure, rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
success in placing feeding tube

SECONDARY OUTCOMES:
- rate of reaching nutritional goal, aspiration pneumonia, feeding tolerance, and pre-albumin

CONTACTS AND LOCATIONS:
Overall Officials: Paul Marik, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital - MRICU, Philadelphia, Pennsylvania, United States